CLINICAL TRIAL: NCT04345965
Title: Sirolimus Eluting Balloon Utilization for Treatment of Vasculogenic Erectile Dysfunction - The SUASION Study
Brief Title: Sirolimus Eluting Balloon Utilization for Treatment of Vasculogenic Erectile Dysfunction
Acronym: SUASION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica San Gaudenzio (Other)
Responsible Party: Principal Investigator, Giuseppe Sangiorgi, Professor, Clinica San Gaudenzio
Other Study IDs: SUASION
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction | interventions — Endovascular Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active endovascular treatment: Patients with erectile dysfunction (ED) and no-response to phosphodiesterase-5 inhibitors for at least 6 months before enrollment
  Interventions: Procedure: Endovascular procedure

INTERVENTIONS:
Procedure: Endovascular procedure — Endovascular therapies for erectile dysfunction

SUMMARY:
Brief Summary:

Background and pathophysiology: Erectile dysfunction (ED) is defined as the recurrent inability to achieve and maintain an erection satisfactory for sexual intercourse.

ED is not in itself a "serious" disease, but its impact on quality of life is extremely important, affecting the family and interpersonal relationships.

Male erection is a complex mechanism that involves neuro-vascular tissue responses with several phases including arterial dilatation, smooth muscle cells relaxation and ultimately veno-occlusive activation.

Vasculogenic erectile dysfunction can be divided in arteriogenic (when there is insufficiency of arterial component of erection due to atherosclerotic plaque encroachment of the penile arteries) or venogenic (where there is insufficiency of the venous component of erection for venous endoleak) Standard treatment Erectile dysfunction is commonly treated by oral phosphodiesterase-5-inhibitor (PDE5i) administration. However, up to 50% of men have a suboptimal response to PDE5-i therapy with the need of additional therapies. New treatment Only recently several studies have been published on percutaneous treatment of ED using plain old balloon angioplasty (POBA), Drug eluting balloons (both paclitaxel and sirolimus, PEB and SES) and drug eluting stents (DES).

Aim of the study: Evaluation of the safety and feasibility of sirolimus drug eluting balloon treatment in focal atherosclerotic lesions of the internal pudendal arteries among men with erectile dysfunction (ED) and a no response to phosphodiesterase-5 inhibitors.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is defined as the recurrent inability to achieve and maintain an erection satisfactory for sexual intercourse ED is not in itself a "serious" disease, but its impact on quality of life is extremely important, affecting the family and interpersonal relationships. Depression, shame, decreased self-esteem and relationship problems are commonly reported symptoms and experiences to people suffering from ED.

Therefore, successful treatment of ED has a strong impact on quality of life. More than 150 million men worldwide have ED, and 52% of men in the United States 40 to 70 years of age report some degree of ED.

The male erection is a complex mechanism that involves neuro-vascular-tissue responses. In particular, the erection mechanism includes a phase of arterial dilation, the relaxation of the musculature of the trabecular smooth muscle cells at the level of the cavernous bodies and, ultimately, the activation of a veno-occlusive at the level of the same mechanism.

Restoring adequate arterial inflow in patients with penile arterial insufficiency can improve erectile function. Surgical re-vascularization has been used successfully in younger men after blunt perineal trauma or pelvic fracture. Older subjects can have obstructive atherosclerotic disease identified by angiography in the iliac, internal pudendal, and cavernosal arteries. Although endovascular revascularization with balloon angioplasty has resulted in at least short-term improvement of erectile function, there have been no prior reports on the feasibility of Sirolimus eluting balloon treatment for ED.

ED counts various causes including psychological factors, neurological hormonal, iatrogenic and to particular lifestyle. A careful collection of the clinical history is essential to identify risk factors for ED: present diseases, drug therapies, previous surgery, smoking and use of drugs.

Clinical examination should aim to assess the secondary sexual characteristics, size and consistency of the testes, perianal sensation, tone of the anal sphincter associated to digital rectal examination and the bulb-cavernous reflection. Palpation of the penis is important to detect the presence of penile plaques indicative of induration penis plastica (Peyronie's disease) and the digital rectal examination provides an opportunity to perform a prostate exam.

The cardiovascular examination should include, in addition to measuring blood pressure and heart rate, the evaluation of peripheral arterial pulses. It has been shown that a good anamnestic collection and a correct clinical examination have a sensitivity of 95% (specificity but much less: about 50%) for a diagnosis of ED of organic origin. For this reason, a definitive diagnosis also requires a diagnostic-instrumental study and laboratory Drug Eluting Balloons (DEBs) represent an attractive and novel treatment modality that offers numerous theoretical advantages over standard angioplasty and stent technologies. Among these benefits: homogenous distribution of an anti-proliferative drug to the vessel wall (not just to segments of the wall in direct contact with stent struts); immediate drug release without the use of a polymer that could trigger late thrombosis; no prolonged, direct drug contact with the arterial wall, allowing better re-endothelialization of the vessel if a bare metal stent (BMS) is used in conjunction; no foreign object left in the body, which is especially important in peripheral applications where stents have been used with suboptimal results; maintenance of original vessel anatomy and flexibility, important during superficial femoral artery re-vascularization especially; and finally, lower restenosis rates in some indications.

The objective of this study is to evaluate of the safety and feasibility of sirolimus drug eluting balloon treatment in focal atherosclerotic lesions of the internal pudendal arteries among men with erectile dysfunction (ED) and no-response to phosphodiesterase-5 inhibitors for at least 6 months before enrollment.

Currently available Drug Coated Balloons (DCBs) in the market are Paclitaxel Eluting Balloon (PEB) - in which paclitaxel is delivered using various drug carriers - and, very recently, Sirolimus Eluting Balloon (SEB). Paclitaxel is cytotoxic drug and can lead to toxicity whereas cytostatic properties of Limus drugs not prone to toxicity as safety margin of sirolimus is higher multiple-folds compared to paclitaxel.

However, due to lipophilic properties of Sirolimus, short term delivery of the drug is thought to be a major challenge. Recently, nanotechnology has being applied to drug eluting balloon. Nanotechnology may offer the advantages of a larger surface area, higher bio-availability, less dose, higher in tissue uptake, and finally good adhesion properties on balloon. With this technology, sirolimus delivery from balloon has been reported to be successful.

Magic Touch™ is a sirolimus nanocarrier coated balloon catheter currently approved for coronary use in Europe. Nanocarriers of sirolimus are encapsulated with a unique phospholipid drug carrier. The drug dose is 180 µg on 3.00 X 15mm (1.27 µg/mm2). The drug carrier has unique cell mimicking properties as well as a phospholipid bi-layer allowing drug retention at higher levels even at very low dose of sirolimus.

This is an observational, retrospective-prospective multicenter registry in patients evaluating the use of Sirolimus Eluting Balloon for the treatment of de novo stenosis in native internal pudendal arteries.

The study population will include 100 patients (10% estimated dropout) affected by vasculogenic ED non responder to PDE5i with up to 2 de novo atherosclerotic artery lesions requiring treatment.

After visual examination, the device must be selected in accordance with the instruction for use (IFU), provided with the device.

The total population in this study will be 100 patients. All patients who meet all the eligibility criteria will be asked to participate. This study will be conducted as a retrospective-prospective "hybrid" study. Two different and specific informed consent forms are provided for patients to be enrolled.

* Prospective patients are informed of the objectives of the study and what their participation in the study will entail.
* Retrospective-prospective patients already underwent angioplasty with the DCB in study consistently with all the eligibility criteria will be informed that their participation will involve the collection of data on their previous angioplasty and participation in the follow-up visits foreseen by the protocol.

Once the patient's eligibility has been determined and the attending physician agrees, a member of the Research Team will approach the patient to initiate the informed consent process The background of the proposed study and the benefits and risks of the procedures and of the study will be explained to the patient.

In both forms the patient is informed that his private data will be protected in accordance with current legislation. The patient must sign the informed consent form prior to enrolment. Failure to obtain a signed informed consent renders the patient ineligible for the study.

ELIGIBILITY:
* Male able to understand and sign a witnessed informed consent for the procedure
* Age >18 years
* Eligibility for percutaneous peripheral intervention
* Patients with ED evaluated by International Index of Erectile Function- (IIEF)-5 score < 15, positive dynamic doppler (PSV <25 cm/sec) and/or evidence at basal CT angiography of single or multiple atherosclerotic lesions in the pudendal arteries
* Hemodynamic conditions must be stable (systolic BP > 100 heart rate (HR) > 40 < 100).
* Left ventricular ejection fraction (LVEF) ≥40% as measured prior to enrollment.
* No response to any dosage of PDE5i for more than 6 mos before enrollment (either chronic or on-demanding).

Angiographic inclusion criteria

* Target lesions must be de novo lesions located in at least one native pudendal artery with a visually estimated reference vessel diameter (RVD) 1.5 mm and 2.5 mm.
* If two lesions in the same vessel are treated, overlapping balloon treatment is allowed.
* Target lesion must be in the pudendal arteries or dorsalis penis with visually estimated stenosis >70% and <100%.

Exclusion Criteria:

* Ejection Fraction below 40%
* Hemodynamic instability (systolic blood pressure <100 mm Hg; heart rate <40 bpm or >100 bpm; complex ventricular arrhythmias; AtrioVentricular (AV) block) requiring balloon counterpulsation or inotropic support.
* Patient was never treated with PDE5i
* Patient has not performed a basal and dynamic pelvic Doppler
* Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Patient has a white blood cell (WBC) count <3,000 cells/mm3
* Patient is on dialysis or has known renal insufficiency (serum creatinine > 2 mg/dl, or Glomerular Filtration Rate (GFR) <40)
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Patient has a known allergy to Sirolimus or protocol required concomitant medications (clopidogrel, thienopyridines, aspirin, contrast) that cannot be adequately premedicated
* Patient has an active peptic ulcer or active gastrointestinal (GI) bleeding
* Patient has a history of coagulopathy
* Patient has other serious medical illness (eg, cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
* Patient is participating in another investigational drug or device clinical trial that has not reached its primary endpoint

Angiographic exclusion criteria

* Vessel size < 1.5 mm by visual estimation.
* Lesion length > 80 mm by visual estimation.
* Restenosis from previous intervention
* Thrombus, or possible thrombus, present in the target vessel
* Previous implantation of a bare/DES in the target vessel

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with erectile dysfunction (ED) and no-response to phosphodiesterase-5 inhibitors for at least 6 months before enrollment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Delta International Index of Erectile Function IEF-5 score between basal and 8 months FU (>5) | 1-8 months
  The score 22-25 means normal function The score 17-21 means very light erectile disfunction The score 12-16 means light to moderate erectile disfunction The score 8-11 means moderate erectile disfunction The score 5-7 means severe erectile disfunction Delta PSV (>8) at the Dynamic Doppler evaluation between basal and 8 mos follow-up

SECONDARY OUTCOMES:
Number of participants Reporting Any Medically Attended Adverse Events (MAEs) | 1-24 months
  The rate of MAE through 1 to 24 months during follow-up evaluated as rate of Death, myocardial infarction (MI), Stroke cases during follow-up.
  In particular:
  * Number of subjects died during follow-up
  * Number of subjects reporting Myocardial Infarction (MI) during follow-up
  * Number of subjects reporting Stroke during follow-up
The rate of Binary Restenosis | 1, 6, 12, 24 months
  Binary restenosis (defined as 50% or greater diameter stenosis in a previously successfully treated lesion as demonstrated by angiographic imaging) in patients who will repeat control angiography if clinically indicated for ED recurrence (clinically evaluated by either needs to reintroduce/increase phosphodiesterase 5 inhibitors (PDEF5i) dosage on- demand), or in patients with bilateral disease with scheduled procedure after 6 mos FU from the index procedure.
Angiographic in-stent late loss measure | 1, 6, 12, 24 months
  Angiographic in-stent late loss measure (where In-stent late loss was defined as the difference between minimum lumen diameter immediately after implantation and that obtained at angiographic follow-up) in patients who will repeat control angiography if clinically indicated for ED recurrence (clinically evaluated by either needs to reintroduce/increase phosphodiesterase 5 inhibitors (PDEF5i) dosage on- demand), or in patients with bilateral disease with scheduled procedure after 6 mos FU from the index procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangiorgi G, Colantonio R, Antonini G, Savino A, Sperandio M. [Percutaneous intervention therapy for vascular erectile dysfunction]. G Ital Cardiol (Rome). 2016 Oct;17(10 Suppl 1):12S-21. doi: 10.1714/2372.25474. Italian. PMID 27729664
- [Background] Diehm N, Marggi S, Ueki Y, Schumacher D, Keo HH, Regli C, Do DD, Moeltgen T, Grimsehl P, Wyler S, Schoenhofen H, Raber L, Schumacher M. Endovascular Therapy for Erectile Dysfunction-Who Benefits Most? Insights From a Single-Center Experience. J Endovasc Ther. 2019 Apr;26(2):181-190. doi: 10.1177/1526602819829903. Epub 2019 Feb 11. PMID 30741067
- [Background] McCabe MP, Sharlip ID, Atalla E, Balon R, Fisher AD, Laumann E, Lee SW, Lewis R, Segraves RT. Definitions of Sexual Dysfunctions in Women and Men: A Consensus Statement From the Fourth International Consultation on Sexual Medicine 2015. J Sex Med. 2016 Feb;13(2):135-43. doi: 10.1016/j.jsxm.2015.12.019. PMID 26953828
- [Background] Johannes CB, Araujo AB, Feldman HA, Derby CA, Kleinman KP, McKinlay JB. Incidence of erectile dysfunction in men 40 to 69 years old: longitudinal results from the Massachusetts male aging study. J Urol. 2000 Feb;163(2):460-3. PMID 10647654
- [Background] Brotons FB, Campos JC, Gonzalez-Correales R, Martin-Morales A, Moncada I, Pomerol JM. Core document on erectile dysfunction: key aspects in the care of a patient with erectile dysfunction. Int J Impot Res. 2004 Oct;16 Suppl 2:S26-39. doi: 10.1038/sj.ijir.3901240. PMID 15496854
- [Background] Lue TF. Erectile dysfunction. N Engl J Med. 2000 Jun 15;342(24):1802-13. doi: 10.1056/NEJM200006153422407. No abstract available. PMID 10853004
- [Background] Ayta IA, McKinlay JB, Krane RJ. The likely worldwide increase in erectile dysfunction between 1995 and 2025 and some possible policy consequences. BJU Int. 1999 Jul;84(1):50-6. doi: 10.1046/j.1464-410x.1999.00142.x. PMID 10444124
- [Background] Gratzke C, Angulo J, Chitaley K, Dai YT, Kim NN, Paick JS, Simonsen U, Uckert S, Wespes E, Andersson KE, Lue TF, Stief CG. Anatomy, physiology, and pathophysiology of erectile dysfunction. J Sex Med. 2010 Jan;7(1 Pt 2):445-75. doi: 10.1111/j.1743-6109.2009.01624.x. PMID 20092448
- [Background] Lue TF. Physiology of penile erection and pathophysiology of erectile dysfunction. In: Saunders W, editor Campbell-Walsh Urology. Philadelphia, 2012.
- [Background] Lue TF, Tanagho EA. Physiology of erection and pharmacological management of impotence. J Urol. 1987 May;137(5):829-36. doi: 10.1016/s0022-5347(17)44267-4. No abstract available. PMID 3553617
- [Background] Kumar V. The Relationship between lipid profile and hypertension. J Med Sci Clin Res 2018;5:40-44.
- [Background] Koncz L, Balodimos MC. Impotence in diabetes mellitus. Med Times. 1970 Aug;98(8):159-70. No abstract available. PMID 5454743
- [Background] Herman A, Adar R, Rubinstein Z. Vascular lesions associated with impotence in diabetic and nondiabetic arterial occlusive disease. Diabetes. 1978 Oct;27(10):975-81. doi: 10.2337/diab.27.10.975. PMID 700261
- [Background] Gupta BP, Murad MH, Clifton MM, Prokop L, Nehra A, Kopecky SL. The effect of lifestyle modification and cardiovascular risk factor reduction on erectile dysfunction: a systematic review and meta-analysis. Arch Intern Med. 2011 Nov 14;171(20):1797-803. doi: 10.1001/archinternmed.2011.440. Epub 2011 Sep 12. PMID 21911624
- [Background] Giuliano FA, Leriche A, Jaudinot EO, de Gendre AS. Prevalence of erectile dysfunction among 7689 patients with diabetes or hypertension, or both. Urology. 2004 Dec;64(6):1196-201. doi: 10.1016/j.urology.2004.08.059. PMID 15596196
- [Background] Angelini G, Pezzini F, Mucci P. [Arteriosclerosis and impotence]. Minerva Psichiatr. 1985 Oct-Dec;26(4):353-17. No abstract available. Italian. PMID 4094548
- [Background] Araujo AB, Hall SA, Ganz P, Chiu GR, Rosen RC, Kupelian V, Travison TG, McKinlay JB. Does erectile dysfunction contribute to cardiovascular disease risk prediction beyond the Framingham risk score? J Am Coll Cardiol. 2010 Jan 26;55(4):350-6. doi: 10.1016/j.jacc.2009.08.058. PMID 20117441
- [Background] Bhatt DL, Steg PG, Ohman EM, Hirsch AT, Ikeda Y, Mas JL, Goto S, Liau CS, Richard AJ, Rother J, Wilson PW; REACH Registry Investigators. International prevalence, recognition, and treatment of cardiovascular risk factors in outpatients with atherothrombosis. JAMA. 2006 Jan 11;295(2):180-9. doi: 10.1001/jama.295.2.180. PMID 16403930
- [Background] Billups KL, Bank AJ, Padma-Nathan H, Katz S, Williams R. Erectile dysfunction is a marker for cardiovascular disease: results of the minority health institute expert advisory panel. J Sex Med. 2005 Jan;2(1):40-50; discussion 50-2. doi: 10.1111/j.1743-6109.2005.20104_1.x. PMID 16422903
- [Background] Dong JY, Zhang YH, Qin LQ. Erectile dysfunction and risk of cardiovascular disease: meta-analysis of prospective cohort studies. J Am Coll Cardiol. 2011 Sep 20;58(13):1378-85. doi: 10.1016/j.jacc.2011.06.024. PMID 21920268
- [Background] Marma AK, Berry JD, Ning H, Persell SD, Lloyd-Jones DM. Distribution of 10-year and lifetime predicted risks for cardiovascular disease in US adults: findings from the National Health and Nutrition Examination Survey 2003 to 2006. Circ Cardiovasc Qual Outcomes. 2010 Jan;3(1):8-14. doi: 10.1161/CIRCOUTCOMES.109.869727. Epub 2009 Nov 16. PMID 20123666
- [Background] Hauri D. Penile revascularization surgery in erectile dysfunction. Urol Int. 2003;70(2):132-40. doi: 10.1159/000068187. PMID 12592042
- [Background] Ginestie J, Romieu A. [The treatment of impotence of vascular origin. Revascularisation of the corpora cavernosa]. J Urol Nephrol (Paris). 1976 Oct-Nov;82(10-11):853-9. French. PMID 1003600
- [Background] Goldwasser B, Carson CC 3rd, Braun SD, McCann RL. Impotence due to the pelvic steal syndrome: treatment by iliac transluminal angioplasty. J Urol. 1985 May;133(5):860-1. doi: 10.1016/s0022-5347(17)49258-5. No abstract available. PMID 3157806
- [Background] Gray RR, Keresteci AG, St Louis EL, Grosman H, Jewett MA, Rankin JT, Provan JL. Investigation of impotence by internal pudendal angiography: experience with 73 cases. Radiology. 1982 Sep;144(4):773-80. doi: 10.1148/radiology.144.4.7111723.
- [Background] Braun M, Wassmer G, Klotz T, Reifenrath B, Mathers M, Engelmann U. Epidemiology of erectile dysfunction: results of the 'Cologne Male Survey'. Int J Impot Res. 2000 Dec;12(6):305-11. doi: 10.1038/sj.ijir.3900622. PMID 11416833
- [Background] Moreira ED Jr, Lbo CF, Diament A, Nicolosi A, Glasser DB. Incidence of erectile dysfunction in men 40 to 69 years old: results from a population-based cohort study in Brazil. Urology. 2003 Feb;61(2):431-6. doi: 10.1016/s0090-4295(02)02158-1. PMID 12597962
- [Background] Schouten BW, Bosch JL, Bernsen RM, Blanker MH, Thomas S, Bohnen AM. Incidence rates of erectile dysfunction in the Dutch general population. Effects of definition, clinical relevance and duration of follow-up in the Krimpen Study. Int J Impot Res. 2005 Jan-Feb;17(1):58-62. doi: 10.1038/sj.ijir.3901264. PMID 15510192
- [Background] Parazzini F, Menchini Fabris F, Bortolotti A, Calabro A, Chatenoud L, Colli E, Landoni M, Lavezzari M, Turchi P, Sessa A, Mirone V. Frequency and determinants of erectile dysfunction in Italy. Eur Urol. 2000 Jan;37(1):43-9. doi: 10.1159/000020098. PMID 10671784
- [Background] Gazzaruso C, Giordanetti S, De Amici E, Bertone G, Falcone C, Geroldi D, Fratino P, Solerte SB, Garzaniti A. Relationship between erectile dysfunction and silent myocardial ischemia in apparently uncomplicated type 2 diabetic patients. Circulation. 2004 Jul 6;110(1):22-6. doi: 10.1161/01.CIR.0000133278.81226.C9. Epub 2004 Jun 21. PMID 15210604
- [Background] Rosen R, Altwein J, Boyle P, Kirby RS, Lukacs B, Meuleman E, O'Leary MP, Puppo P, Robertson C, Giuliano F. Lower urinary tract symptoms and male sexual dysfunction: the multinational survey of the aging male (MSAM-7). Eur Urol. 2003 Dec;44(6):637-49. doi: 10.1016/j.eururo.2003.08.015. PMID 14644114
- [Background] Rosen MP, Greenfield AJ, Walker TG, Grant P, Dubrow J, Bettmann MA, Fried LE, Goldstein I. Cigarette smoking: an independent risk factor for atherosclerosis in the hypogastric-cavernous arterial bed of men with arteriogenic impotence. J Urol. 1991 Apr;145(4):759-63. doi: 10.1016/s0022-5347(17)38444-6. PMID 2005695
- [Background] De Angelis L, Marfella MA, Siniscalchi M, Marino L, Nappo F, Giugliano F, De Lucia D, Giugliano D. Erectile and endothelial dysfunction in Type II diabetes: a possible link. Diabetologia. 2001 Sep;44(9):1155-60. doi: 10.1007/s001250100616. PMID 11596671
- [Background] Montorsi P, Ravagnani PM, Galli S, Rotatori F, Veglia F, Briganti A, Salonia A, Deho F, Rigatti P, Montorsi F, Fiorentini C. Association between erectile dysfunction and coronary artery disease. Role of coronary clinical presentation and extent of coronary vessels involvement: the COBRA trial. Eur Heart J. 2006 Nov;27(22):2632-9. doi: 10.1093/eurheartj/ehl142. Epub 2006 Jul 19. PMID 16854949
- [Background] Vlachopoulos C, Jackson G, Stefanadis C, Montorsi P. Erectile dysfunction in the cardiovascular patient. Eur Heart J. 2013 Jul;34(27):2034-46. doi: 10.1093/eurheartj/eht112. Epub 2013 Apr 24. PMID 23616415
- [Background] Shamloul R, Ghanem H. Erectile dysfunction. Lancet. 2013 Jan 12;381(9861):153-65. doi: 10.1016/S0140-6736(12)60520-0. Epub 2012 Oct 5. PMID 23040455
- [Background] Gandaglia G, Briganti A, Jackson G, Kloner RA, Montorsi F, Montorsi P, Vlachopoulos C. A systematic review of the association between erectile dysfunction and cardiovascular disease. Eur Urol. 2014 May;65(5):968-78. doi: 10.1016/j.eururo.2013.08.023. Epub 2013 Aug 23. PMID 24011423
- [Background] Philip F, Shishehbor MH, Desai MY, Schoenhagen P, Ellis S, Kapadia SR. Characterization of internal pudendal artery atherosclerosis using aortography and multi-detector computed angiography. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):E516-21. doi: 10.1002/ccd.24804. Epub 2013 Apr 16. PMID 23553996
- [Background] Shishehbor MH, Philip F. Endovascular treatment for erectile dysfunction: an old paradigm revisited. J Am Coll Cardiol. 2012 Dec 25;60(25):2628-30. doi: 10.1016/j.jacc.2012.09.032. Epub 2012 Nov 21. No abstract available. PMID 23177299
- [Background] Thompson IM, Tangen CM, Goodman PJ, Probstfield JL, Moinpour CM, Coltman CA. Erectile dysfunction and subsequent cardiovascular disease. JAMA. 2005 Dec 21;294(23):2996-3002. doi: 10.1001/jama.294.23.2996. PMID 16414947
- [Background] Montorsi F, Briganti A, Salonia A, Rigatti P, Margonato A, Macchi A, Galli S, Ravagnani PM, Montorsi P. Erectile dysfunction prevalence, time of onset and association with risk factors in 300 consecutive patients with acute chest pain and angiographically documented coronary artery disease. Eur Urol. 2003 Sep;44(3):360-4; discussion 364-5. doi: 10.1016/s0302-2838(03)00305-1. PMID 12932937
- [Background] Hodges LD, Kirby M, Solanki J, O'Donnell J, Brodie DA. The temporal relationship between erectile dysfunction and cardiovascular disease. Int J Clin Pract. 2007 Dec;61(12):2019-25. doi: 10.1111/j.1742-1241.2007.01629.x. PMID 17997808
- [Background] Solomon H, Man JW, Wierzbicki AS, Jackson G. Relation of erectile dysfunction to angiographic coronary artery disease. Am J Cardiol. 2003 Jan 15;91(2):230-1. doi: 10.1016/s0002-9149(02)03113-2. No abstract available. PMID 12521639
- [Background] Castaneda-Zuniga WR, Smith A, Kaye K, Rusnak B, Herrerra M, Miller R, Amplatz K, Weens C, Ketchum D. Transluminal angioplasty for treatment of vasculogenic impotence. AJR Am J Roentgenol. 1982 Aug;139(2):371-3. doi: 10.2214/ajr.139.2.371. No abstract available. PMID 6211967
- [Background] Dewar ML, Blundell PE, Lidstone D, Herba MJ, Chiu RC. Effects of abdominal aneurysmectomy, aortoiliac bypass grafting and angioplasty on male sexual potency: a prospective study. Can J Surg. 1985 Mar;28(2):154-6, 159. PMID 3155988
- [Background] Hall SA, Shackelton R, Rosen RC, Araujo AB. Sexual activity, erectile dysfunction, and incident cardiovascular events. Am J Cardiol. 2010 Jan 15;105(2):192-7. doi: 10.1016/j.amjcard.2009.08.671. PMID 20102917
- [Background] Rogers JH, Goldstein I, Kandzari DE, Kohler TS, Stinis CT, Wagner PJ, Popma JJ, Jaff MR, Rocha-Singh KJ. Zotarolimus-eluting peripheral stents for the treatment of erectile dysfunction in subjects with suboptimal response to phosphodiesterase-5 inhibitors. J Am Coll Cardiol. 2012 Dec 25;60(25):2618-27. doi: 10.1016/j.jacc.2012.08.1016. Epub 2012 Nov 21. PMID 23177300
- [Background] Salem S, Abdi S, Mehrsai A, Saboury B, Saraji A, Shokohideh V, Pourmand G. Erectile dysfunction severity as a risk predictor for coronary artery disease. J Sex Med. 2009 Dec;6(12):3425-32. doi: 10.1111/j.1743-6109.2009.01515.x. Epub 2009 Sep 30. PMID 19796020
- [Background] Urigo F, Pischedda A, Maiore M, Salis A, Picciau M, Carboni M, Conti M, Canalis GC. [Role of arteriography and percutaneous transluminal angioplasty in the diagnosis and treatment of arterial vasculogenic impotence]. Radiol Med. 1994 Jul-Aug;88(1-2):86-92. Italian. PMID 8066261
- [Background] Van Unnik JG, Marsman JW. Impotence due to the external iliac steal syndrome treated by percutaneous transluminal angioplasty. J Urol. 1984 Mar;131(3):544-5. doi: 10.1016/s0022-5347(17)50490-5. PMID 6230464
- [Background] Wang T, Lee W, Chen W, Chen M. Comprehensive assessment of prevalence and distribution of obstructive pelvic arterial lesions by computed tomographic angiography in patients with erectile dysfunction. American College of Cardiology. San Francisco: Elsevier, 2013:B160.
- [Background] Wang TD, Lee WJ, Yang SC, Lin PC, Tai HC, Hsieh JT, Liu SP, Huang CH, Chen WJ, Chen MF. Safety and six-month durability of angioplasty for isolated penile artery stenoses in patients with erectile dysfunction: a first-in-man study. EuroIntervention. 2014 May;10(1):147-56. doi: 10.4244/EIJV10I1A23. PMID 24832642
- [Background] Cremers B, Speck U, Kaufels N, Mahnkopf D, Kuhler M, Bohm M, Scheller B. Drug-eluting balloon: very short-term exposure and overlapping. Thromb Haemost. 2009 Jan;101(1):201-6. PMID 19132209
- [Background] Radke PW, Joner M, Joost A, Byrne RA, Hartwig S, Bayer G, Steigerwald K, Wittchow E. Vascular effects of paclitaxel following drug-eluting balloon angioplasty in a porcine coronary model: the importance of excipients. EuroIntervention. 2011 Oct 30;7(6):730-7. doi: 10.4244/EIJV7I6A116. PMID 21986331
- [Background] Takimura CK, Galon MZ, Gutierrez PS, Sojitra P, Vyas A, Doshi M, Lemos PA. A new polymer-free drug-eluting stent with nanocarriers eluting sirolimus from stent-plus-balloon compared with bare-metal stent and with biolimus A9 eluting stent in porcine coronary arteries. Cardiovasc Diagn Ther. 2015 Apr;5(2):113-21. doi: 10.3978/j.issn.2223-3652.2015.03.08. PMID 25984451
- [Background] Lemos PA, Farooq V, Takimura CK, Gutierrez PS, Virmani R, Kolodgie F, Christians U, Kharlamov A, Doshi M, Sojitra P, van Beusekom HM, Serruys PW. Emerging technologies: polymer-free phospholipid encapsulated sirolimus nanocarriers for the controlled release of drug from a stent-plus-balloon or a stand-alone balloon catheter. EuroIntervention. 2013 May 20;9(1):148-56. doi: 10.4244/EIJV9I1A21. PMID 23685303
- [Background] Parikh KH, Shetty R, Dani S, Bhatt P, Doshi M-, Sojitra P. Real-world safety and outcome measures of novel sirolimus coated balloon catheter. J Am Coll Cardiol 2016;67:225.
- [Background] Valji K, Bookstein JJ. Transluminal angioplasty in the treatment of arteriogenic impotence. Cardiovasc Intervent Radiol. 1988 Aug;11(4):245-52. doi: 10.1007/BF02577011. PMID 2975966
- [Background] Bahren W, Gall H, Scherb W, Stief C, Thon W. Arterial anatomy and arteriographic diagnosis of arteriogenic impotence. Cardiovasc Intervent Radiol. 1988 Aug;11(4):195-210. doi: 10.1007/BF02577004. PMID 3147134
- [Background] Wang TD, Lee WJ, Yang SC, Lin PC, Tai HC, Liu SP, Huang CH, Chen WJ, Chen MF, Hsieh JT. Clinical and Imaging Outcomes up to 1 Year Following Balloon Angioplasty for Isolated Penile Artery Stenoses in Patients With Erectile Dysfunction: The PERFECT-2 Study. J Endovasc Ther. 2016 Dec;23(6):867-877. doi: 10.1177/1526602816669337. Epub 2016 Sep 14. PMID 27629440
- [Background] Siroky MB, Azadzoi KM. Vasculogenic erectile dysfunction: newer therapeutic strategies. J Urol. 2003 Aug;170(2 Pt 2):S24-9; discussion S29-30. doi: 10.1097/01.ju.0000075361.35942.17. PMID 12853769